CLINICAL TRIAL: NCT02843295
Title: Catalytic Antibodies to Predict Uninvasively Late Transplant Failure
Acronym: CATAPULT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2009-592
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Renal Transplantation
Keywords: renal transplantation; immunology; rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Population of the study (Experimental): 3 stratification groups: Group 1: High immunologic risk Patients receiving a ≥ 2nd graft and/or Panel Reactive Antibody ≥ 30% and/or Human Leukocyte Antigen (HLA) mismatches ≥ 4 Group 2: High non-immunologic risk Donors over 60 years of age and/or Donor between 50 to 59 years of age who have died of stroke, or had a history of high blood pressure, or at the time of death had a creatininemia ≥ 135 µmol/L Group 3: Low risk Patients not included in Groups 1 or 2
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples

SUMMARY:
Chronic Allograft Nephropathy (CAN), a major cause of late allograft failure, is characterized by a progressive decline in graft function correlating with tissue destruction. Recent data suggest that it may be possible to delay graft destruction if adequate management is initiated early (ie, at the stage of subclinical CAN). It is therefore essential to design new tests allowing physicians to predict transplant recipients prone to develop CAN

DETAILED DESCRIPTION:
Superantibodies are multifunctional antibodies combining the classical antigen-binding function with nonclassical biological activities, such as protease-like activity. In the past few years the role of proteolytic SuperAntibody (pSAb) has been evidenced in many biological processes in which their role may be either deleterious (autoimmune disease, alloimmune response against) or beneficial (sepsis).

Nothing is known so far regarding the role of pSAb in the setting of solid organ transplantation.

Preliminary data

The investigator has obtained preliminary results from a retrospective case control study indicating that an elevated serine protease activity of circulating IgG (measured by the hydrolysis of a synthetic fluorescent substrate: Proline-Phenylalanine-Arginine-Methylcoumarinamide (PFR-MCA)), correlates with the absence of CAN on protocol biopsy performed 2 years post-transplantation. Interestingly, low level of proteolysis IgG, measured 3 months post-transplantation, were also predictive of CAN at 2 years down the lane.

Aim of the Research project:

The aim is to validate in a prospective study, the potential of pSAb as predictive marker for CAN

100 recipients of a renal graft have to be enrolled and followed for 2 years.

The level of PFR-MCA hydrolysis by circulating Immunoglobulin G (IgG) will be measured before the transplantation and every 3 months up to one year and every 6 months thereafter until 2 year post-transplantation. The development of CAN will be assessed by estimated glomerular filtration rate (Modification of the Diet in Renal Disease (MDRD) formula), the proteinuria and the histological examination of the graft (screening biopsy at 3 months and 1 year will be analysed using a computerized color image analysis to quantify interstitial fibrosis).

The capacity of the pSAb test to predict CAN will be validated and the sensibility and specificity of this test will be calculated. The optimal cut-off value will be determined from the Receiver Operating Characteristic (ROC) analysis. The accuracy of the test will be evaluated in subgroups displaying various risk factors for CAN.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 the day of transplantation
* Recipient of a renal graft
* Informed consent to participate to the study
* Patient transplanted and followed 2 years in one of the 3 transplantation centers of the study (Hospital Edouard Herriot or Centre Hospitalier Lyon Sud)

Exclusion Criteria:

* Multiorgan transplantation
* Previous transplantation
* ABO incompatible renal transplantation
* Patient > 18 years old but under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
PFR-MCA hydrolysis by circulating IgG (mmol/min/mol) | at 3 months post-transplantation
PFR-MCA hydrolysis by circulating IgG (mmol/min/mol) | at 6 months post-transplantation
PFR-MCA hydrolysis by circulating IgG (mmol/min/mol) | at 9 months post-transplantation
PFR-MCA hydrolysis by circulating IgG (mmol/min/mol) | at 12 months post-transplantation
PFR-MCA hydrolysis by circulating IgG (mmol/min/mol) | at 18 months post-transplantation
PFR-MCA hydrolysis by circulating IgG (mmol/min/mol) | at 24 months post-transplantation

SECONDARY OUTCOMES:
Glomerular filtration rate by MDRD formula (ml/min) | at 3 months post-transplantation
Glomerular filtration rate by MDRD formula (ml/min) | at 6 months post-transplantation
Glomerular filtration rate by MDRD formula (ml/min) | at 9 months post-transplantation
Glomerular filtration rate by MDRD formula (ml/min) | at 12 months post-transplantation
Glomerular filtration rate by MDRD formula (ml/min) | at 18 months post-transplantation
Glomerular filtration rate by MDRD formula (ml/min) | at 24 months post-transplantation
Proteinuria/creatinuria ratio (g/g) | at 3 months post-transplantation
Proteinuria/creatinuria ratio (g/g) | at 6 months post-transplantation
Proteinuria/creatinuria ratio (g/g) | at 9 months post-transplantation
Proteinuria/creatinuria ratio (g/g) | at 12 months post-transplantation
Proteinuria/creatinuria ratio (g/g) | at 18 months post-transplantation
Proteinuria/creatinuria ratio (g/g) | at 24 months post-transplantation
Interstitial fibrosis on graft biopsy (%) | at day 0
Interstitial fibrosis on graft biopsy (%) | at 12 months post-transplantation
Interstitial fibrosis on graft biopsy (%) | at 24 months post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Olivier THAUNAT, MD, Principal Investigator — Hospices Civils de Lyon - Transplantation Department
Locations (1):
- Transplantation Department, Lyon, France

IPD SHARING:
Plan to Share IPD: No